CLINICAL TRIAL: NCT01823133
Title: A Randomized, Open Label Crossover Study to Investigate the Pharmacokinetic Drug Interactions Between Gemigliptin and Rosuvastatin in Healthy Male Subjects
Brief Title: Study for Investigate the Pharmacokinetic Drug Interactions Between Gemigliptin and Rosuvastatin
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: LG Life Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: LG-GSCL001
Record Dates: First submitted 2013-03-28; First posted 2013-04-04 (Estimated); Last update posted 2013-08-28 (Estimated); Status verified 2013-08

CONDITIONS: Healthy
MeSH Terms: interventions — LC15-0444; Rosuvastatin Calcium

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- gemigliptin only (Experimental): Multiple administrations of gemigliptin
  Interventions: Drug: gemigliptin only
- rosuvastatin only (Experimental): Multiple administrations of rosuvastatin
  Interventions: Drug: rosuvastatin only
- gemigliptin and rosuvastatin (Experimental): Multiple administrations of gemigliptin and rosuvastatin
  Interventions: Drug: gemigliptin and rosuvastatin

INTERVENTIONS:
Drug: gemigliptin only — gemigliptin 50mg qd on day 1~7
  Arms: gemigliptin only
Drug: rosuvastatin only — rosuvastatin 20mg qd on day 1~7
  Arms: rosuvastatin only
Drug: gemigliptin and rosuvastatin — gemigliptin 50mg, rosuvastatin 20mg qd on day 1~7
  Arms: gemigliptin and rosuvastatin

SUMMARY:
Investigate the pharmacokinetic drug interactions between gemigliptin and rosuvastatin in healthy subjects

ELIGIBILITY:
Inclusion Criteria:

* Age between 20 to 45, healthy male subjects (at screening)
* BMI between 18 - 27 kg/m2 (at screening)
* Blood pressure SBP 90-140 mmHg, DBP 60-95 mmHg
* FPG 70-125mg/dL glucose level (at screening)
* Subject who totally understand the progress of this clinical trials, make decision by his free will, and signed a consent form to follow the

Exclusion Criteria:

* Subject who has past or present history of any diseases following below.(liver including hepatitis virus carrier, kidney, Neurology,immunology,pulmonary,endocrine,hematooncology,cardiology,mental disorder.)
* Subject who had GI tract disease that influencable to drug absorption or(ulcer, acute or chronic pancreatitis) surgery.(appendectomy, hernioplasty are not included)
* Subject who had drug hypersensitivity reaction.(gemigliptin, rosuvastatin, aspirin, antibiotics)
* Subject who already admitted in other investigator product in 80 days
* Subject who had whole blood donation in 60 days, or component blood donation in 30 days or transfusion in 30 days currently

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2013-04; Primary Completion 2013-05 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Cmax | up to 72 hour post dose
  to evaluate Cmax of gemigliptin and rosuvastatin at steady state
AUC | up to 72 hour post dose
  to evaluate AUCt of gemiglipin, rosuvastatin, and metabolite LC15-0636, N-desmethylrosuvastatin at steady state

SECONDARY OUTCOMES:
Tmax | up to 72 hour post dose
  to evaluate time of Cmax at steady state, gemiglipin, rosuvastatin, and metabolite LC15-0636, N-desmethylrosuvastatin
Cmin | upto 72 hour post dose
  to evaluate Cmin of gemigliptin and rosuvastatin at steady state
t1/2β | upto 72 hour post dose
  to evaluate half-life of gemiglipin, rosuvastatin, and metabolite LC15-0636, N-desmethylrosuvastatin
Cmax | upto 72 hour post dose
  to evaluate Cmax of metabolite LC15-0636, N-desmethylrosuvastatin at steady state
AUC | upto 72 hour post dose
  to evaluate AUC of metabolite LC15-0636, N-desmethylrosuvastatin at steady state
metabolic ratio | upto 72 hour post dose
  to evaluate metabolic ratio of gemiglipin and rosuvastatin

CONTACTS AND LOCATIONS:
Locations (1):
- Asan Medical Center, Seoul, South Korea

REFERENCES:
- [Derived] Choi HY, Lim HS, Kim YH, Jeon HS, Kim MJ, Lee SH, Jung JH, Lee YK, Kim HJ, Bae KS. Evaluation of the pharmacokinetics of the DPP-4 inhibitor gemigliptin when coadministered with rosuvastatin or irbesartan to healthy subjects. Curr Med Res Opin. 2015 Feb;31(2):229-41. doi: 10.1185/03007995.2014.980886. Epub 2014 Nov 6. PMID 25350224